CLINICAL TRIAL: NCT05862532
Title: TeTrimTeas: Gut Microbiome and Blood Lipid Markers After Habitual Herbal Tea Consumption
Brief Title: Gut Microbiome and Blood Markers After Habitual Herbal Tea Consumption
Acronym: SRTT
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aberystwyth University (Other)
Collaborators: TeTrimTeas Cyf (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 23306
Record Dates: First submitted 2023-04-24; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-04

CONDITIONS: Obesity; Well-being
Keywords: Herbal tea infusions; Lipid composition; Gut microbiome; Short Chain fatty acids; Well-being
MeSH Terms: conditions — Obesity | interventions — Sennosides; Tea

STUDY DESIGN:
Intervention Model Description: Two intervention arms and one placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Welsh Herbal tea with Senna (Experimental): Welsh Herbal tea with green tea and Senna
  Interventions: Dietary Supplement: TeTrimTeas welsh Herbal tea with senna
- Welsh Herbal tea with rhubarb root (Experimental): Welsh Herbal tea with green tea and rhubarb root
  Interventions: Dietary Supplement: TeTrimTeas welsh Herbal tea with rhubarb root
- Green tea (Active Comparator): Dartmoor green tea
  Interventions: Dietary Supplement: TeTrimTeas welsh Herbal tea with green tea

INTERVENTIONS:
Dietary Supplement: TeTrimTeas welsh Herbal tea with rhubarb root — TeTrimTeas welsh Herbal tea with green tea and rhubarb root
  Arms: Welsh Herbal tea with rhubarb root
Dietary Supplement: TeTrimTeas welsh Herbal tea with senna — TeTrimTeas welsh Herbal tea with green tea and senna
  Arms: Welsh Herbal tea with Senna
Dietary Supplement: TeTrimTeas welsh Herbal tea with green tea — TeTrimTeas welsh Herbal tea with green tea
  Arms: Green tea

SUMMARY:
TeTrimTeas intends is to establish a long-term cooperative with local growers and producers who will become partners in the business, with profit share to local growers and producers. The overall aim of the company is to produce quality, science-based botanical/herbal teas to improve health and wellbeing, growing as many of the ingredients locally and organically, to reduce food-to-fork miles within the decarbonisation and sustainability agendas in Wales.

TeTrimTeas have created herbal green tea blends, improving on existing Chinese formulation, and would like to test it as 'health tea'. The recruited cohort will be randomised into one of three intervention teas (green tea control, senna herbal mix and rhubarb root herbal mix). They would like to explore if consumption of the teas for 21 days has an impact on digestion and potentially help control weight gain.

Aberystwyth University will use high resolution metabolomics to investigate the chemical composition of capillary blood samples, in particular the short chain fatty acids. They will also assess lipid composition in capillary bloods and the microbiome of stools. Diet data, stool consistency and anthropometric measurements will be collected pre and post intervention. Results will advance product development and data would be used in grant applications into the health benefits of the herbal teas.

DETAILED DESCRIPTION:
TeTrimTeas has created herbal green tea blends, improving on existing Chinese formulation, and would like to test it as 'health tea'. The recruited cohort will be randomised into one of three intervention teas (green tea control, senna herbal mix and rhubarb root herbal mix). This will be double blinded so neither the participant nor the researcher will know what group they have been allocated into. Information can be disclosed at the end of the study. Participants will come to WARU or Trimsaran Community Health Centre for induction and study visits.

The experimental sequence

'Diet-monitoring' period (two days before the study)

Prior to the experimental session it is important that all participants undergo a period where foods are recorded. This will help the researchers interpret any results after consumption of the test/control food. The researchers would ask them to refrain from taking any over-the-counter medication (such as ibuprofen, paracetamol, aspirin, cough/ cold remedies) or herbal supplements, and to let us know if they find that it is necessary to take any such medication during the trial.

Experimental session- 21 days

Morning: Participants will come to WARU or Trimsaran Community Health Centre for their pre-organised timeslot to allow researchers to collect a fasted capillary (fingerpick) blood samples and stool sample. They may consume their breakfast after their visit. They will also collect their tea bags. Researchers will also take participants weight and height and collect diet data (PDQS) and stool scores (Bristol Stool scale).

Over 21 days: the researchers would ask the participants to consume a cup of tea after their last meal/snack of the day (post 6pm) daily, for 21 days. The researchers would ask them not to consume anything after the tea. In a cup/mug the researchers would ask them to place a 2.5g tea bag and add 190ml of hot water (80-100◦C) and stir clockwise 10 consecutive times to allow for optimal infusion and then allow to brew for 5 minutes, before removal.

After the experimental period:

Before their final visit (or at their final visit): the researchers would like participants to fill in another food questionnaire and a stool scale.

Morning of their final visit. The researchers would ask the participant to come to WARU or Trimsaran Community Health Centre for their pre-organised timeslot to allow us to collect a fasted capillary (fingerpick) blood samples and stool sample. The researchers will also take their weight and height. They may consume their breakfast after their visit. Afterwards, they can go back to their 'normal' eating pattern.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adults >18 y Age
* Commit to fasting capillary blood collection
* Commit to stool sampling collection
* Able to refrain from taking any over-the-counter medication or herbal supplements during the diet monitoring and experimental periods.
* Able to prepare and consume the tea during the experimental days, after the last meal/snack of the day and not to consume anything afterwards
* Fill in diet diaries, FFQ and stool ranking
* Able to inform the researcher if any antibiotics or heavy alcohol is consumed over the intervention period

Exclusion Criteria

* Showing (or anyone within the household) any COVID-19 symptoms (see COVID-19 basic health screen)*
* Higher risk or vulnerable from coronavirus or live with someone at a higher risk of a severe illness from COVID-19 (over 70, undergoing cancer treatment, high risk of getting infections).
* Had a letter from the NHS advising you to shield (isolate)
* Had been at risk of exposure to COVID-19 such as travel, contact with someone with COVID-19, been exposed to the virus, or has been asked to self-isolate by the track and trace system.
* Serious health conditions that require daily long-term medications (including immunosuppressants)
* A history or current diabetes, lung issues, gut inflammation (Crohns, IBD), digestive disorders
* Diagnosed with a serious health condition within the last 12 months
* Pregnant
* Play sports at a high level (more than 7h/week or 1h/day)
* Smoking
* consume high dose of alcohol > 21 unit per week for men and > 14 units per week for women
* Food allergy /food intolerance/ eating disorder or are on a specially prescribed diet

  * If the potential participant has had COVID-19 previously (and are fully recovered and not within isolation) then they are eligible to join the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in total plasma Cholesterol after the rhubarb root tea | Decrease from Baseline plasma Cholesterol after 21 days
  Change in total Cholesterol (mmol/L) after the rhubarb root tea measured in capillary bloods using AFINION S100
Change in total plasma Cholesterol after the rhubarb root tea | Decrease from total Cholesterol plasma after the rhubarb root tea when compared with senna tea plasma Cholesterol after 21 days
  Change in total Cholesterol (mmol/L) after the rhubarb root tea measured in capillary bloods using AFINION S100
Change in total plasma Cholesterol after the rhubarb root tea | Decrease from total Cholesterol plasma after the rhubarb root tea when compared with green tea plasma Cholesterol after 21 days
  Change in total Cholesterol (mmol/L) after the rhubarb root tea measured in capillary bloods using AFINION S100
Change in total plasma Cholesterol after the senna tea | Decrease from Baseline plasma Cholesterol after 21 days
  Change in total Cholesterol (mmol/L) after the senna tea measured in capillary bloods using AFINION S100
Change in total plasma Cholesterol after the green tea | Decrease from Baseline plasma Cholesterol after 21 days
  Change in total Cholesterol (mmol/L) after the green tea measured in capillary bloods using AFINION S100
Change in plasma Low density lipoprotein cholesterol (LDL-C) after the rhubarb root tea | Decrease from Baseline plasma Low density lipoprotein cholesterol (LDL-C) after 21 days
  Change in Low density lipoprotein cholesterol (LDL-C) (mmol/L) after the rhubarb root tea measured in capillary bloods using AFINION S100
Change in plasma Low density lipoprotein cholesterol (LDL-C) after the rhubarb root tea | Decrease from plasma Low density lipoprotein cholesterol (LDL-C) after the rhubarb root tea when compared with senna tea plasma Low density lipoprotein cholesterol (LDL-C) after 21 days
  Change in Low density lipoprotein cholesterol (LDL-C) (mmol/L) after the rhubarb root tea measured in capillary bloods using AFINION S100
Change in plasma Low density lipoprotein cholesterol (LDL-C) after the rhubarb root tea | Decrease from plasma Low density lipoprotein cholesterol (LDL-C) after the rhubarb root tea when compared with green tea plasma Low density lipoprotein cholesterol (LDL-C) after 21 days
  Change in Low density lipoprotein cholesterol (LDL-C) (mmol/L) after the rhubarb root tea measured in capillary bloods using AFINION S100
Change in plasma Low density lipoprotein cholesterol (LDL-C) after the senna tea | Decrease from Baseline plasma Low density lipoprotein cholesterol (LDL-C) after 21 days
  Change in Low density lipoprotein cholesterol (LDL-C) (mmol/L) after the senna tea measured in capillary bloods using AFINION S100
Change in plasma Low density lipoprotein cholesterol (LDL-C) after the green tea | Decrease from Baseline plasma Low density lipoprotein cholesterol (LDL-C) after 21 days
  Change in Low density lipoprotein cholesterol (LDL-C) (mmol/L) after the green tea measured in capillary bloods using AFINION S100

SECONDARY OUTCOMES:
Change in plasma High-Density Lipoprotein cholesterol (HDL-C) after the rhubarb root tea | Increase from Baseline plasma High-Density Lipoprotein cholesterol (HDL-C) after 21 days
  Change in High-Density Lipoprotein cholesterol (HDL-C) (mmol/L) after the rhubarb root tea measured in capillary bloods using AFINION S100
Change in plasma High-Density Lipoprotein cholesterol (HDL-C) after the rhubarb root tea | Increase of plasma High-Density Lipoprotein cholesterol (HDL-C) after Rhubarb root tea when compared with senna tea plasma High-Density Lipoprotein cholesterol (HDL-C) after 21 days
  Change in High-Density Lipoprotein cholesterol (HDL-C) (mmol/L) after the rhubarb root tea measured in capillary bloods using AFINION S100
Change in plasma High-Density Lipoprotein cholesterol (HDL-C) after the rhubarb root tea | Increase of plasma High-Density Lipoprotein cholesterol (HDL-C) after Rhubarb root tea when compared with green tea plasma High-Density Lipoprotein cholesterol (HDL-C) after 21 days
  Change in High-Density Lipoprotein cholesterol (HDL-C) (mmol/L) after the rhubarb root tea measured in capillary bloods using AFINION S100
Change in plasma High-Density Lipoprotein cholesterol (HDL-C) after the senna tea | Increase from Baseline plasma High-Density Lipoprotein cholesterol (HDL-C) after 21 days
  Change in High-Density Lipoprotein cholesterol (HDL-C) (mmol/L) after the senna tea measured in capillary bloods using AFINION S100
Change in plasma High-Density Lipoprotein cholesterol (HDL-C) after the green tea | Increase from Baseline plasma High-Density Lipoprotein cholesterol (HDL-C) after 21 days
  Change in High-Density Lipoprotein cholesterol (HDL-C) (mmol/L) after the green tea measured in capillary bloods using AFINION S100
Change in plasma Triglycerides after the rhubarb root tea | Decrease from Baseline plasma Triglycerides after 21 days
  Change in Triglycerides (mmol/L) after the rhubarb root tea measured in capillary bloods using AFINION S100
Change in plasma Triglycerides after the senna tea | Decrease from senna tea plasma Triglycerides after 21 days
  Change in Triglycerides (mmol/L) after the senna measured in capillary bloods using AFINION S100
Change in plasma Triglycerides after the green tea | Decrease from green tea plasma Triglycerides after 21 days
  Change in Triglycerides (mmol/L) after the green tea measured in capillary bloods using AFINION S100
Change in plasma Triglycerides after the rhubarb root tea | Decrease from rhubarb root plasma Triglycerides after 21 days when compared with senna tea plasma Triglycerides after 21 days
  Change in Triglycerides (mmol/L) after the rhubarb root tea measured in capillary bloods using AFINION S100
Change in plasma Triglycerides after the rhubarb root tea | Decrease from rhubarb root plasma Triglycerides after 21 days when compared with green tea plasma Triglycerides after 21 days
  Change in Triglycerides (mmol/L) after the rhubarb root tea measured in capillary bloods using AFINION S100
Change in plasma non- high-density lipoprotein cholesterol (total cholesterol - high-density lipoprotein cholesterol) after the rhubarb root tea | Decrease from Baseline plasma non- high-density lipoprotein cholesterol (total cholesterol - high-density lipoprotein cholesterol) after 21 days
  Change in non- high-density lipoprotein cholesterol (total cholesterol - high-density lipoprotein cholesterol) (mmol/L) after the rhubarb root tea measured in capillary bloods using AFINION S100
Change in plasma non- high-density lipoprotein cholesterol (total cholesterol - high-density lipoprotein cholesterol) after the senna tea | Decrease from senna tea plasma non- high-density lipoprotein cholesterol (total cholesterol - high-density lipoprotein cholesterol) after 21 days
  Change in non- high-density lipoprotein cholesterol (total cholesterol - high-density lipoprotein cholesterol) (mmol/L) after the senna tea measured in capillary bloods using AFINION S100
Change in plasma non- high-density lipoprotein cholesterol (total cholesterol - high-density lipoprotein cholesterol) after the green tea | Decrease from green tea plasma non- high-density lipoprotein cholesterol (total cholesterol - high-density lipoprotein cholesterol) after 21 days
  Change in non- high-density lipoprotein cholesterol (total cholesterol - high-density lipoprotein cholesterol) (mmol/L) after the green tea measured in capillary bloods using AFINION S100
Change in plasma non- high-density lipoprotein cholesterol (total cholesterol - high-density lipoprotein cholesterol) after the rhubarb root tea | Decrease of plasma non- high-density lipoprotein cholesterol (total cholesterol - high-density lipoprotein cholesterol) after 21 days of the rhubarb root tea when compared with 21 days of the senna tea
  Change in non- high-density lipoprotein cholesterol (total cholesterol - high-density lipoprotein cholesterol) (mmol/L) after the after the rhubarb root tea measured in capillary bloods using AFINION S100
Change in plasma non- high-density lipoprotein cholesterol (total cholesterol - high-density lipoprotein cholesterol) after the rhubarb root tea | Decrease of plasma non- high-density lipoprotein cholesterol (total cholesterol - high-density lipoprotein cholesterol) after 21 days of the rhubarb root tea when compared with 21 days of the green tea
  Change in non- high-density lipoprotein cholesterol (total cholesterol - high-density lipoprotein cholesterol) (mmol/L) after the rhubarb root tea measured in capillary bloods using AFINION S100
Diet choices change measured using the Prime Diet Quality Score | Increased score from baseline Prime Diet Quality Score at 21 days after the Rhubarb root tea
  Measured using the Prime Diet Quality Score. The Prime Diet Quality Score (PDQS) measures intake of the 22 component foods/food groups over the last 30 days with seven possible responses for each component ranging from "once a month or less" to "≥ 2 times/day." Scores are then summed to create a PDQS total diet quality score with a possible score from 0 to 126 with higher scores indicating a healthier diet.
Diet choices change measured using the Prime Diet Quality Score | Increased score from baseline Prime Diet Quality Score at 21 days after the senna tea
  Measured using the Prime Diet Quality Score. The Prime Diet Quality Score (PDQS) measures intake of the 22 component foods/food groups over the last 30 days with seven possible responses for each component ranging from "once a month or less" to "≥ 2 times/day." Scores are then summed to create a PDQS total diet quality score with a possible score from 0 to 126 with higher scores indicating a healthier diet.
Diet choices change measured using the Prime Diet Quality Score | Increased score from baseline Prime Diet Quality Score at 21 days after the green tea
  Measured using the Prime Diet Quality Score. The Prime Diet Quality Score (PDQS) measures intake of the 22 component foods/food groups over the last 30 days with seven possible responses for each component ranging from "once a month or less" to "≥ 2 times/day." Scores are then summed to create a PDQS total diet quality score with a possible score from 0 to 126 with higher scores indicating a healthier diet.
Diet choices change measured using the Prime Diet Quality Score | Increased score from the Rhubarb root tea Prime Diet Quality Score at 21 days compared with the senna tea at 21 days
  Measured using the Prime Diet Quality Score. The Prime Diet Quality Score (PDQS) measures intake of the 22 component foods/food groups over the last 30 days with seven possible responses for each component ranging from "once a month or less" to "≥ 2 times/day." Scores are then summed to create a PDQS total diet quality score with a possible score from 0 to 126 with higher scores indicating a healthier diet.
Diet choices change measured using the Prime Diet Quality Score | Increased score from the Rhubarb root tea Prime Diet Quality Score at 21 days compared with the green tea at 21 days
  Measured using the Prime Diet Quality Score. The Prime Diet Quality Score (PDQS) measures intake of the 22 component foods/food groups over the last 30 days with seven possible responses for each component ranging from "once a month or less" to "≥ 2 times/day." Scores are then summed to create a PDQS total diet quality score with a possible score from 0 to 126 with higher scores indicating a healthier diet.
BMI change measured by weight and height | Decrease score from baseline BMI Score at 21 days after the Rhubarb root tea
  BMI change measured by weight and height will be combined to report BMI in kg/m^2
BMI change measured by weight and height | Decrease score from baseline BMI Score at 21 days after the senna tea
  BMI change measured by weight and height will be combined to report BMI in kg/m^2
BMI change measured by weight and height | Decrease score from baseline BMI Score at 21 days after the green tea
  BMI change measured by weight and height will be combined to report BMI in kg/m^2
BMI change measured by weight and height | Decreased score from the Rhubarb root tea BMI at 21 days compared with the senna tea at 21 days
  BMI change measured by weight and height will be combined to report BMI in kg/m^2
BMI change measured by weight and height | Decreased score from the Rhubarb root tea BMI at 21 days compared with the green tea at 21 days
  BMI change measured by weight and height will be combined to report BMI in kg/m^2
Changes in short chain fatty acids concentrations in plasma | Increased concentration of total short chain fatty acids from baseline concentration at 21 days after the Rhubarb root tea
  Changes in short chain fatty acids concentrations in plasma measured using Gas Chromatography-Flame Ionization Detection
Changes in short chain fatty acids concentrations in plasma | Increased concentration of total short chain fatty acids from baseline concentration at 21 days after the senna tea
  Changes in short chain fatty acids concentrations in plasma measured using Gas Chromatography-Flame Ionization Detection
Changes in short chain fatty acids concentrations in plasma | Increased concentration of total short chain fatty acids from baseline concentration at 21 days after the green tea
  Changes in short chain fatty acids concentrations in plasma measured using Gas Chromatography-Flame Ionization Detection
Changes in short chain fatty acids concentrations in plasma | Increased concentration of total short chain fatty acids after the rhubarb root tea at 21 days compared with the senna tea after 21 days
  Changes in short chain fatty acids concentrations in plasma measured using Gas Chromatography-Flame Ionization Detection
Changes in short chain fatty acids concentrations in plasma | Increased concentration of total short chain fatty acids after the rhubarb root tea at 21 days compared with the green tea after 21 days
  Changes in short chain fatty acids concentrations in plasma measured using Gas Chromatography-Flame Ionization Detection

CONTACTS AND LOCATIONS:
Locations (1):
- Well-being and Health Assessment Research Unit (WARU), Aberystwyth, Ceredigion, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be available to other researchers.

DOCUMENTS (1):
  • Study Protocol (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/32/NCT05862532/Prot_000.pdf